CLINICAL TRIAL: NCT02941692
Title: The Effects of Oxytocin on Couples Conflict Resolution Interactions
Brief Title: Oxytocin for Couples Conflict Resolution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 31736; K12HD055885 (NIH)
Record Dates: First submitted 2015-10-01; First posted 2016-10-21 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Substance Misuse; Interpersonal Conflict; Neuroendocrine Reactivity
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): Participants randomized to this condition will receive 40 IU dose of intranasal oxytocin.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Participants randomized to this condition will receive a matching dose of intranasal saline spray as placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Placebo — Placebo for Oxytocin
  Arms: Placebo

SUMMARY:
Oxytocin is a promising new medication found to have positive effects on prosocial behavior, reduce negative affect such as fear and anxiety, and reduce stress-induced addictive behaviors. This study aims to investigate the extent to which a 40 IU dose of intranasal oxytocin improves couples' conflict resolution skills and subjective, physiological, and neuroendocrine responses to conflict. Conflict resolution discussions will take place in the laboratory and will be videotaped.

DETAILED DESCRIPTION:
Substance use disorders (SUD) are characterized by dysregulation of the hypothalamic-pituitary axis (HPA). The neuropeptide oxytocin, commonly administered as an intranasal spray, is a drug that has prominent anxiolytic and prosocial effects on human behaviors. While the mechanisms of action facilitating the behavioral effects of oxytocin in humans is complex and many questions about this process remain, there is a consensus in the existing literature that oxytocin modulates HPA axis reactivity to stressful social stimuli. Preliminary studies suggest that oxytocin is known to reduce couple conflict among normative couples. A more developed line of research indicates that oxytocin mitigates addictive behaviors in the context of various drugs of abuse. Given the high prevalence and severity of dyadic conflict among couples where one or both partner has substance abuse, and given the salience of dyadic conflict as a precipitant to substance use behaviors, it is critical to investigate the therapeutic effects of oxytocin among couples with substance use problems. Namely, oxytocin holds promise as a potential augmenter for conjoint couples therapies, particularly those targeting the reduction of substance use problems. However, only two studies have examined the effects of oxytocin on couples' communication behaviors. Those two studies found that couples' communication skills improved following the administration of oxytocin. It is important to extend this line of research to examine conflict resolution skills among couples with substance use problems. To date, no studies have examined the effects of oxytocin on subjective, physiological, or neuroendocrine reactivity to dyadic conflict. The present study aims to fill that gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. both partners are willing to participate, and
3. at least one partner has engaged in hazardous drinking (i.e. 4 or more drinks for women, 6 or more for men) or illicit drug use during the past 60 days

Exclusion Criteria:

1. pregnancy for women
2. current psychotic or bipolar disorders
3. active suicidal or homicidal ideation and intent
4. subjects who would present a serious suicide risk, such as those with severe depression, or who are likely to require hospitalization during the course of the study
5. severe, unilateral intimate partner violence in the past year
6. BMI greater than 39.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxytocin: Participants randomized to this condition will receive 40 IU dose of intranasal oxytocin.
  Oxytocin
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 32 | 34
Completed | 32 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.97 (10.17) | 32.21 (9.73) | 32.08 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two same-sex couples were excluded from analyses to accommodate multi-level modeling approach. one couple was excluded from analyses due to questionable reliability of data.
  Participants
    Female | 16 | 14 | 30
    Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two same-sex couples were excluded from analyses to accommodate multilevel modeling analyses. One couple was excluded from analyses due to unreliability of data.
  Participants
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 17 | 14 | 31
    White | 13 | 11 | 24
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Distress Maintaining Attributions
Description: Couples' conflict resolution discussions are video recorded and coded according to an observational coding system: the Rapid Marital Interaction Coding System, which assesses the frequency of behaviors (distress maintaining attributions and relationship enhancing attributions) during the 10 minute conflict resolution discussion. This variable is operationalized as the number of instances of distress maintaining attributions during each of two ten minute conflict resolution discussions.
Time Frame: Frequency of distress maintaining attrbibutions per 10 minutes
Population: Analyses were limited to heterosexual couples with reliable data reporting in order to accommodate the data analytic approach (i.e., multilevel modeling).
Measure: Mean (Standard Deviation); unit: distress maintaining attributions
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 32 | 28
distress maintaining attributions | .81 (2.67) | -.48 (2.51)

2. Secondary Outcome: Change in Salivary Cortisol (μg/dL)
Description: Cortisol samples are collected at baseline, pre-post each conflict resolution discussion, and at 15, 30, and 60 minute post-task intervals.
Time Frame: Measured at 7 time points: Baseline, immediately before and after Conflict Resolution Task #1, Immediately after Conflict Resolution Task #2, and at 15, 30, and 60 minutes following the completion of Conflict Resolution task #2.
Population: Three couples (6 total participants) were not included in analyses.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 28 | 32
μg/dL
  Time 1 (Baseline) | .28 (.18) | .30 (.20)
  Time 2 (Pre Conflict Discussion #1) | .25 (.14) | .29 (.18)
  Time 3 (Post Conflict Discussion #1) | .18 (.11) | .21 (.12)
  Time 4 (Post Conflit Discussion #2) | .17 (.11) | .22 (.16)
  Time 5 (15 minutes Post Conflict Discussion) | .16 (.10) | .22 (.20)
  Time 6 (30 minutes Post Conflict Discussion) | .17 (.10) | .22 (.18)
  Time 7 (60 Minutes Post Conflict Discussion) | .16 (.08) | .19 (.13)

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Description: This study employed the same adverse event definition as clinicaltrials.gov
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 0/32 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT02941692/Prot_SAP_000.pdf